CLINICAL TRIAL: NCT06971263
Title: Influence of Dietary and Palliative Care Consultation on the Quality of Life (Qol), Performance Status, and Nutritional Status of Cancer Patients in Bangladesh
Acronym: Consult Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jahangirnagar University (Other)
Collaborators: Bangladesh University Grants Commission (UGC) (Unknown)
Responsible Party: Principal Investigator, Syed Billal Hossain, PhD Student, Jahangirnagar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BBEC-JU-M2025-02-199
Record Dates: First submitted 2025-04-17; First posted 2025-05-14 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: Cancer; Dietary Consultation; Palliative Care; Quality of Life; Performance Status; Nutritional Status
MeSH Terms: conditions — Neoplasms | interventions — Palliative Care; Diet, Healthy

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial (RCT)
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Data collectors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cancer patients with both face-to face nutrition and palliative care counselling (Active Comparator): Recruited cancer patients will be given both nutrition and palliative care counselling during face-to face surveys.
  Interventions: Behavioral: Consultation on both nutrition, and palliative care
- Cancer patients with face-to face nutrition counselling (Active Comparator): Recruited cancer patients will be given nutrition counselling on healthy diet during face-to face surveys.
  Interventions: Behavioral: Counselling on nutrition and healthy diet
- Cancer patients without any consultation or intervention (No Intervention): Recruited cancer patients will not be given any nutrition and palliative care counselling or interventions during face-to face surveys.

INTERVENTIONS:
Behavioral: Consultation on both nutrition, and palliative care — The intervention on the nutrition and palliative care components will include open-ended consultations based on ESPEN practical guidelines on nutrition in cancer patients with one cancer center dietitian and one palliative care physician to discuss patient needs and required to improve their health consequences.
  Arms: Cancer patients with both face-to face nutrition and palliative care counselling
Behavioral: Counselling on nutrition and healthy diet — The intervention on the nutrition and healthy diet components will include open-ended consultations based on ESPEN practical guidelines on nutrition in cancer patients with one cancer center dietitian to discuss patient dietary needs for improving their health consequences.
  Arms: Cancer patients with face-to face nutrition counselling

SUMMARY:
Cancer patients are more likely to have malnutrition, which has been associated with poorer quality of life, higher morbidity, mortality rates, and impaired efficacy and tolerance to therapy. Malnutrition is thought to afflict the cancer patients, with weight loss and varied degrees of asthenia being the main symptoms. In fact, malnutrition can increase the risk of surgical complications such as anastomosis dehiscence, poor wound healing, morbidity, and mortality. Quality of Life is among the most important health issues for cancer patients. Patients view it as a specific and complex type of patient-reported outcomes (PROs) that considers their social, economic, psychological, and physical activities. The quality of life for cancer patients is often lower than for the general population. Despite the fact that several studies in the Western population have suggested a relationship between nutritional status and quality of life (QoL). There aren't many reliable, in-depth studies on the effectiveness of nutritional testing and early malnutrition therapy, as well as to look at the nutritional health and quality of life of cancer patients in Bangladesh. Therefore, the aim of this study is to outline the Influence of Dietary and Palliative Care Consultation on the Quality of Life (Qol), Performance Status, and Nutritional Status of Cancer Patients in Bangladesh. To conduct this randomized control trial (RCT), data will be collected through 3 observations: baseline survey with two follow-up surveys on the following months from the selected cohorts of cancer patients who will be receiving cancer treatments. There will be two groups of cohort, one will be given nutrition and palliative care counselling will be given as intervention during each observation and another group will be without consultancy. "The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire version 3.0 (EORTC-QLQ C30)", "The Patient-Generated Subjective Global Assessment PG-SGA)" to estimate nutritional status, and "The Eastern Cooperative Oncology Group's (ECOG) scale" to determine the performance status (PS) will be used as instruments to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Cancer Patients under standard treatment, Willing to participate, Who can eat orally, and Health indicators are measurable.

Exclusion Criteria:

* Cancer Patients under no standard treatment, Not willing to participate, Who cannot eat orally, Health indicators are not measurable, and Death.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Patient-Generated Subjective Global Assessment (PG-SGA) Scale | From enrollment to the end of interventions at 10 weeks.
  The Patient-Generated Subjective Global Assessment (PG-SGA) instrument will be used to diagnose nutrition. The technique permits categorizing the nutritional evaluation into three groups: A for well-nourished, B for suspected or moderate malnutrition, and C for severe malnutrition. Weight in kilograms divided by height in squared meter is known as the body mass index (BMI). In addition to PG-SGA, BMI will be calculated and categorized according to the age-specific and sex-specific chart created by the US Centers for Disease Control and Prevention.

SECONDARY OUTCOMES:
Eastern Cooperative Oncology Group's (ECOG) scale | From enrollment to the end of interventions at 10 weeks.
  The Eastern Cooperative Oncology Group's (ECOG) scale will be used to determine the performance status (PS). The ECOG divides performance scales into five categories: "Zero- fully active"; "One -limited in physically demanding activity but ambulatory and able to perform work of a light or sedentary nature"; "Two- refers to being ambulatory and capable of all self-care but unable to perform any work activities"; "Three- limited capacity for self- care"; "Four- refers to being completely inactive"; and "Five- Dead".

OTHER OUTCOMES:
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire version 3.0 (EORTC-QLQ-C30) scale | From enrollment to the end of interventions at 10 weeks.
  The EORTC-QLQ-C30 will be used in all patients to assess Quality of Life. This instrument is a 30-item cancer-specific questionnaire including six function scales (physical, emotional, cognitive, social, role, and global health/QoL), three symptom scales (fatigue, pain, nausea/ vomiting), and six single items assessing symptoms and the financial impact of the disease. Higher scores on the function scales indicate better functioning whilst higher scores on the symptom scales and single items denote increased symptomatology or worse financial impairment. Original scores will be linearly transformed to obtain quantified scores within the range 0 to 100. In addition, for better validation in the clinical context, overall scores derived from function scales, symptom scales and single items, will be calculated on the basis of the very high statistical significance of inter-scale correlations according to to EORTC's guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Billal Hossain, MPH, Principal Investigator — Jahangirnagar University
Locations (3):
- Bangladesh (3):
  - Chittagong Medical College Hospital (CMCH), Chittagong, Chattogram
  - Department of Public Health and Informatics, Jahangirnagar University, Savar Upazila, Dhaka Division
  - Mymensingh Medical College Hospital (MMCH), Mymensingh, Mymensingh

IPD SHARING:
Plan to Share IPD: Yes
IPD related to the cancer patients with intervention might be shared on reasonable requests related to research, review and citation.
Supporting Information: Study Protocol, ICF
Time Frame: April 2026 to March 2028
Access Criteria: Access to IPD will be given on reasonable requests related to research, review and citation.

REFERENCES:
- See also: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) — https://qol.eortc.org/questionnaire/eortc-qlq-c30/
- See also: Patient-Generated Subjective Global Assessment (PG-SGA) Nutrition scale — https://pt-global.org/pt-global/
- See also: Eastern Cooperative Oncology Group's (ECOG) Performance Status scale — https://ecog-acrin.org/resources/ecog-performance-status/